CLINICAL TRIAL: NCT03543904
Title: Effects of Pre- Operative Physiotherapy Education and Post Operative Physiotherapy in Children With Abdominal Surgery
Brief Title: Pre-operative and Post-operative Physiotherapy in Children With Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor and Research Scholar, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDU/IEC/1189; U1111-1213-2267 (Registry Identifier: Universal Trial Number (UTN)); L-79385/2018 (Other: Copyright office, Government of India)
Record Dates: First submitted 2018-05-05; First posted 2018-06-01 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Abdominal Surgery
Keywords: Abdomen; Children; Chest physical therapy; Surgery

STUDY DESIGN:
Intervention Model Description: Parallel
Masking Description: Participants were blinded towards which group they were allocated. If participants know that they were belonging to the experimental group 1 then they will be performing better than the participants in allocated in the experimental group 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-operative physiotherapy education (Experimental): Pre-operative education regarding post-operative physiotherapy intervention and post-operative physiotherapy intervention in children with abdominal surgery
  Interventions: Procedure: Pre-operative physiotherapy education; Procedure: Post-operative physiotherapy intervention
- Post-OP PT without Pre-OP education (Experimental): Post-operative physiotherapy intervention without pre-operative education in children with abdominal surgery
  Interventions: Procedure: Post-operative physiotherapy intervention

INTERVENTIONS:
Procedure: Pre-operative physiotherapy education — Pre-operative education regarding post-operative physiotherapy intervention in children with abdominal surgery which includes,
  1. Deep breathing exercises
  2. Pursed lip breathing exercises
  3. Diaphragmatic breathing exercises
  4. Leg ROM (active hip and knee flexion, extension and abduction exercises)
  5. Ankle toe movements exercises
  Arms: Pre-operative physiotherapy education
Procedure: Post-operative physiotherapy intervention — Post-operative physiotherapy intervention which includes,
  1. Deep breathing exercises
  2. Pursed lip breathing exercises
  3. Diaphragmatic breathing exercises
  4. Leg ROM (active hip and knee flexion, extension and abduction exercises)
  5. Ankle toe movements exercises

SUMMARY:
The study will be conducted in a pediatric surgery ward, department of pediatrics. Children between the ages of 5 to 17 years who underwent for abdominal surgery will be recruited by simple random sampling. Parents of all the potential participants will receive a written explanation of the trial and given written informed consent forms to be signed prior to their child being involved in the trial. Pre- op physiotherapy education is given to one experimental group and after surgery post operative treatment is given to both the experimental groups. spirometery, 6 minute walk test, 10 meter walk test, Timed up and go test and Nine star stair climbing test will be used for data collection.

DETAILED DESCRIPTION:
Pre- operative education is given to the experimental group 1 only. Pre- op. physiotherapy education includes-

Pursed lip breathing exercises × 10 repetitions Diaphragmatic breathing exercises × 10 repetitions Leg ROM (active hip and knee flexion, extension and abduction exercises) and ankle toe movements exercises × 10 repititions

Post- op. physiotherapy will be given to both the experimental groups. it includes- On Post operative day 1

Deep breathing exercises- Pursed lip breathing exercises × Diaphragmatic breathing exercises (5 repetitions × 2 sets)

Segmental breathing exercises × 5 repetitions × 2 sets Incentive spirometer 10 breaths up to 600 cc (In three sets) per session Leg Range of motion exercises (active hip and knee flexion and extension exercises) × 5 repetitions × 2 sets Ankle and toe movements× 10 repetitions × 2 sets Ambulation program High sitting minimum of 2 min Static March for 1 min Walk for 5 min. every 2 hourly

Post operative day 2 Deep breathing exercises- Pursed lip breathing exercises × Diaphragmatic breathing exercises (5 repetitions × 2 sets) Segmental breathing exercises × 5 repetitions × 2 sets Incentive spirometer 10 breaths upto 600 cc (In three sets) per sessionThoracic expansion exercises- ACBT (Active cycles of breathing techniques)

Diaphragmatic breathing (10 rep.), deep breathing (5 sec. hold), huffing x 2 repetitions twice a day Walk for 10 min. every 2 hourly

Post operative day 3 Pursed lip breathing exercises x 10 repetitions x 2 sets Incentive spirometer 10 breaths upto 900cc (In three sets) per session Thoracic expansion exercises- ACBT Diaphragmatic breathing (5-10 rep.), deep breathing (5 sec. hold), huffing x 2 repetitions twice a day Walk for 15 min. every 2 hourly

Post operative day 4 Incentive spirometer/ 10breaths upto 900cc (In three sets) per session Walk for 20 min. every 4 hourly

Post operative day 5 Incentive spirometer / 10breaths upto 1000cc (In three sets) per session Stair climbing up to 9 steps in ascending and descending pattern for 5 minutes rest in between

ELIGIBILITY:
Inclusion Criteria:

* Children having following abdominal incision- inguinal incision, left subcostal incision, right subcostal incision, kehr incision, McBurney incision, Transverse incison, thoraco-abdominal incison, Median and paramedian incision12
* Between ages of 5 to 17 years
* Who follows and obeys the commands
* Children who is willing to participate in the study

Exclusion Criteria:

* Children who requires organ transplants
* With mental retardation
* With physical disability

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
Change in FVC (Liters) (spirometric measurements) | 3 times (recorded pre operative and post operative on day1 and 5)
  Functional vital capacity (FVC) is the maximum volume of air which can be exhaled or inspired during a forced maneuver

SECONDARY OUTCOMES:
6 minute walk test | 2 times (recorded pre operative and post operative on day 5)
  the child will be asked to walk far as possible for 6 minutes. Child will be encouraged in every minute for walking. At 6 minute, child will be asked to stop. If the participant stops at any time prior record the distance at which the oxygen saturation drops < 88%
10 meter walk test | 3 times (recorded pre operative and post operative on day1 and 5)
  The 10MWT assesses walking speed in meters per second over a short duration.The child will be asked to walk a set distance (10 meters). Time will be measured during walking. The distance covered is divided by the time it took the individual to walk that distance.
Nine stair climbing test | 2 times (recorded pre operative and post operative on day 5)
  It is performed for measuring functional strength and balance through ascending and descending a set number of steps. 2min. time will be given to complete the test. The patient should use the assistive device (if any) normally used to perform the activity at the time of testing.
Timed up and go test | 3 times (recorded pre operative and post operative on day1 and 5)
  The child starts in a seated position. The child will be tands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the child is seated.

OTHER OUTCOMES:
Change in FEV1 (Liters) (Spirometeric measurements) | 3 times (recorded pre operative and post operative on day1 and 5)
  Forced expiratory volume in the first second (FEV1) Is the volume expired in the first second of maximal expiration after a full inspiration
Change in FEV1/ FVC (%) (Spirometric measurements) | 2 times (recorded pre operative and post operative on day 5)
  It is also known as Tiffeneau pinelli index (FEV1/FVC) represents the proportion of individual's vital capacity that they are able to expire in the first second of forced expiration to full, forced vital capacity
Change in PEFR (Liters) [Peak Expiratory Flow Rate (liters)] (Spirometeric measurements) | 3 times (recorded pre oprative and post operative on day1 and 5)
  Inspiratory vital capacity (IVC) is the maximum volume of air inhaled from the point of maximum expiration
Chest expansion test | 3 times (recorded pre operative and post operative on day1 and 5)
  Chest expansion test measures the expansion of chest when the subject takes a deep breath. Chest expansion will be measured at 3 different levels. i.e 1.) Axillary level 2) Nipple level 3) xiphi-sternum level

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, BPT, MPT, Principal Investigator — Maharishi Markandeshwar institute of physiotherapy and Rehabilitation, MM(DU); Satya Sree, MS, MCh, Study Director — HOD, Department of Pediatric surgery, MMIMSR, MM(DU), Mullana, Haryana
Locations (1):
- Pediatric surgery ward, Maharishi Markandeshwar Hospital, Mullana, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
by Publication in Mendeley Data set
Time Frame: 13 May, 2019 to ever
Access Criteria: Sharma, Neha; Samuel, Asir John (2019), "Effect of Pre-operative physiotherapy education and Post-operative physiotherapy in children with abdominal surgery", Mendeley Data, v1 http://dx.doi.org/10.17632/skkt9tsjd3.1
URL: http://dx.doi.org/10.17632/skkt9tsjd3.1

REFERENCES:
- [Background] Boden I, Skinner EH, Browning L, Reeve J, Anderson L, Hill C, Robertson IK, Story D, Denehy L. Preoperative physiotherapy for the prevention of respiratory complications after upper abdominal surgery: pragmatic, double blinded, multicentre randomised controlled trial. BMJ. 2018 Jan 24;360:j5916. doi: 10.1136/bmj.j5916. PMID 29367198
- [Background] Soares SM, Nucci LB, da Silva MM, Campacci TC. Pulmonary function and physical performance outcomes with preoperative physical therapy in upper abdominal surgery: a randomized controlled trial. Clin Rehabil. 2013 Jul;27(7):616-27. doi: 10.1177/0269215512471063. Epub 2013 Feb 12. PMID 23405020
- [Background] Boden I, Browning L, Skinner EH, Reeve J, El-Ansary D, Robertson IK, Denehy L. The LIPPSMAck POP (Lung Infection Prevention Post Surgery - Major Abdominal - with Pre-Operative Physiotherapy) trial: study protocol for a multi-centre randomised controlled trial. Trials. 2015 Dec 15;16:573. doi: 10.1186/s13063-015-1090-6. PMID 26666321
- [Background] Katsura M, Kuriyama A, Takeshima T, Fukuhara S, Furukawa TA. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD010356. doi: 10.1002/14651858.CD010356.pub2. PMID 26436600
- See also: Preserving pulmonary function and functional capacity in children undergoing open abdominal surgery: A one group pretest-posttest, quasiexperimental pilot trial — http://doi.org/10.1016/j.jpedsurg.2019.10.058
- Available data/document: Pilot study — http://doi.org/10.1016/j.jpedsurg.2019.10.058 — Preserving pulmonary function and functional capacity in children undergoing open abdominal surgery: A one group pretest-posttest, quasiexperimental pilot trial
- Available data/document: Individual Participant Data Set: Version 1 — http://dx.doi.org/10.17632/skkt9tsjd3.1 — Effect of Pre-operative physiotherapy education and Post-operative physiotherapy in children with abdominal surgery", Mendeley Data, v1 http://dx.doi.org/10.17632/skkt9tsjd3.1
- Available data/document: Clinical Study Report — http://doi.org/10.1016/j.jpedsurg.2020.04.007 — A randomized clinical trial in improving pulmonary function and functional capacity in paediatric open abdominal surgery